CLINICAL TRIAL: NCT01774344
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Phase III Study of Regorafenib in Patients With Hepatocellular Carcinoma (HCC) After Sorafenib
Brief Title: Study of Regorafenib After Sorafenib in Patients With Hepatocellular Carcinoma
Acronym: RESORCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15982; 2012-003649-14 (EudraCT Number)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Regorafenib; BAY73-4506
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regorafenib (Experimental): 160 mg orally (p.o.) every day (qd) for 3 weeks of every 4 week cycle (i.e. 3 weeks on, 1 week off) plus BSC (Best Supportive Care)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Placebo (Placebo Comparator): 4 matching placebo tablets for 3 weeks of every 4 week cycle (i.e. 3 weeks on, 1 week off) plus BSC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib, 40 mg tablets
  Arms: Regorafenib
Drug: Placebo — Placebo tablets matching in appearance
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate efficacy and safety of regorafenib in patients with advanced liver cancer who had progressed after sorafenib treatment. Patients were treated with regorafenib or placebo using a 2:1 randomization scheme.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of HCC (hepatocellular carcinoma) or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases criteria in patients with a confirmed diagnosis of cirrhosis
* Barcelona Clinic Liver Cancer stage Category B or C that cannot benefit from treatments of established efficacy with higher priority such as resection, local ablation, chemoembolization or systemic sorafenib.
* Failure to prior treatment with sorafenib (defined as documented radiological progression according to the radiology charter). Randomization needs to be performed within 10 weeks after the last treatment with sorafenib.
* Tolerability of prior treatment with sorafenib defined as not less than 20 days at a minimum daily dose of 400 mg QD within the last 28 days prior to withdrawal.
* Liver function status Child-Pugh Class A. Child Pugh status should be calculated based on clinical findings and laboratory results during the screening period.

Local or loco-regional therapy of intrahepatic tumor lesions (e.g. surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed >/=4 weeks before first dose of study medication. Note: patients who received sole intrahepatic intraarterial chemotherapy, without lipiodol or embolizing agents are not eligible.

* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory tests conducted within 7 days before randomization.
* Glomerular filtration rate >/= 30 ml/min/1.73 m^2 according to the Modification of diet in renal disease study equation.
* At least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST (RECIST version 1.1), and modified RECIST for HCC. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion.
* Life expectancy of at least 3 months.
* Women of childbearing potential and men must agree to use adequate contraception .

Exclusion Criteria :

* Sorafenib treatment within 2 weeks of randomization.
* Prior systemic treatment for HCC, except sorafenib.
* Permanent discontinuation of prior sorafenib therapy due to sorafenib related toxicity.
* Known history or symptomatic metastatic brain or meningeal tumors (head CT or MRI at screening to confirm the absence of central nervous system [CNS] disease if patient has symptoms suggestive or consistent with CNS disease).
* Uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Uncontrolled ascites (defined as not easily controlled with diuretic or paracentesis treatment).
* Ongoing infection > Grade 2 according to NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events) v. 4.0. Hepatitis B is allowed if no active replication is present. Hepatitis C is allowed if no antiviral treatment is required.
* Clinically significant bleeding NCI-CTCAE version 4.0 Grade 3 or higher within 30 days before randomization.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication.
* Patients unable to swallow oral medications.
* Interstitial lung disease with ongoing signs and symptoms at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (128):
- United States (16):
  - Los Angeles, California
  - Orange, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Louisville, Kentucky
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Pittsburgh, Pennsylvania
  - Richmond, Virginia
  - Seattle, Washington
- Pilar, Buenos Aires, Argentina
- Australia (5):
  - Camperdown, New South Wales
  - Liverpool, New South Wales
  - Herston, Queensland
  - Clayton, Victoria
  - Box Hill
- Austria (3):
  - Graz, Styria
  - Linz, Upper Austria
  - Vienna
- Belgium (2):
  - Bruxelles - Brussel
  - La Louvière
- Brazil (2):
  - Salvador, Estado de Bahia
  - São Paulo
- China (16):
  - Hefei, Anhui
  - Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Dalian, Liaoning
  - Xi'an, Shaanxi
  - Chengdu, Sichuan
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Czechia (3):
  - Hradec Králové
  - Olomouc
  - Prague
- France (18):
  - Angers
  - Caen
  - Clichy
  - Créteil
  - Dijon
  - La Tronche
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Perpignan
  - Reims
  - Rennes
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (11):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Hamburg
- Hungary (3):
  - Budapest
  - Debrecen
  - Kaposvár
- Italy (13):
  - Foggia, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Pisa, Tuscany
  - Padua, Veneto
- Japan (12):
  - Chiba, Chiba
  - Kashiwa-shi, Chiba
  - Fukuoka, Fukuoka
  - Iizuka-shi, Fukuoka
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Utsunomiya, Tochigi
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Musashino-shi, Tokyo
- Netherlands (2):
  - Amsterdam
  - Leiden
- Russia (2):
  - Barnaul
  - Moscow
- Singapore, Singapore
- South Korea (3):
  - Busan, Busan Gwang''yeogsi
  - Daegu
  - Seoul
- Spain (6):
  - Oviedo, Principality of Asturias
  - Alicante
  - Barcelona
  - Córdoba
  - Madrid
  - Zaragoza
- Switzerland (2):
  - Bellinzona, Canton Ticino
  - Bern
- Taiwan (3):
  - Kaohsiung City, Kaohsiung
  - Taipei
  - Taoyuan District
- United Kingdom (4):
  - Birmingham, West Midlands
  - Leeds, West Yorkshire
  - Bristol
  - London

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Finn RS, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Gerolami R, Caparello C, Cabrera R, Chang C, Sun W, LeBerre MA, Baumhauer A, Meinhardt G, Bruix J. Outcomes of sequential treatment with sorafenib followed by regorafenib for HCC: Additional analyses from the phase III RESORCE trial. J Hepatol. 2018 Aug;69(2):353-358. doi: 10.1016/j.jhep.2018.04.010. Epub 2018 Apr 26. PMID 29704513
- [Result] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Derived] Wu W, Mao H, Song J, Yang F. Bibliometric analysis of hepatocellular carcinoma and tyrosine kinase inhibitors. Medicine (Baltimore). 2025 May 16;104(20):e42015. doi: 10.1097/MD.0000000000042015. PMID 40388796
- [Derived] Teufel M, Seidel H, Kochert K, Meinhardt G, Finn RS, Llovet JM, Bruix J. Biomarkers Associated With Response to Regorafenib in Patients With Hepatocellular Carcinoma. Gastroenterology. 2019 May;156(6):1731-1741. doi: 10.1053/j.gastro.2019.01.261. Epub 2019 Feb 6. PMID 30738047
- See also: Click here to find information about studies related to Bayer AG products conducted in Europe. — https://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 14 May 2013 (first subject first visit), 29 February 2016 (primary completion date) and 05-July-2019 (Last Patient Last Visit =End of study).
Pre-assignment Details: Overall, 843 subjects were screened, of them 270 subjects were screening failures. 573 subjects were randomized and assigned to treatment; of them 6 subjects never received treatment. 436 Entered survival Follow-up and 4 End of survival follow-up data not available.
Groups:
- Placebo: Subjects received placebo matched to regorafenib coated tablets orally every day for 3 weeks followed by 1 week off treatment plus best best supportive care.
- Regorafenib 160 mg (BAY73-4506): Subjects received regorafenib 160 milligram (mg) (4 * 40 mg coated tablets) orally every day for 3 weeks followed by 1 week off treatment plus BSC.
Period: Overall Study
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Started | 194 | 379
Treated | 193 | 374
Entered Survival FU | 145 | 291
Completed | 132 | 258
Not Completed | 62 | 121
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 4 | 10
Not completed — End of survival follow-up not available | 2 | 2
Not completed — Data collection finished | 4 | 14
Not completed — Other | 0 | 1
Not completed — Did not enter Survival Follow up | 49 | 83

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects received placebo matched to regorafenib coated tablets orally every day for 3 weeks followed by 1 week off treatment plus best supportive care (BSC).
- Total: Total of all reporting groups
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506) | Total
Number analyzed (Participants) | 194 | 379 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.6) | 61.8 (12.4) | 61.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 46 | 69
  Male | 171 | 333 | 504
Eastern cooperative oncology group (ECOG) Performance Status (PS) (data collection system-RAVE) [Count of Participants; unit: Participants] — ECOG PS was measured in a scale from 0 (best) to grade 4 (worst), where 0= Fully active, able to carry on all pre-diseases performance without restriction, 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2= Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50 percent (%) waking hours (h), 3= Capable of only limited self-care, confined to bed/chair, more than 50% waking hours, and 4= Completely disabled, cannot carry on any self-care, totally confined to bed/chair.
  Participants
    ECOG PS 0 | 130 | 247 | 377
    ECOG PS 1 | 64 | 132 | 196
ECOG PS: Interactive voice response system (IVRS) [Count of Participants; unit: Participants] — ECOG PS was measured in a scale from 0 (best) to grade 4 (worst), where 0= Fully active, able to carry on all pre-diseases performance without restriction, 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2= Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50 % waking h, 3= Capable of only limited self-care, confined to bed/chair, more than 50% waking hours, and 4= Completely disabled, cannot carry on any self-care, totally confined to bed/chair.
  Participants
    ECOG PS 0 | 129 | 251 | 380
    ECOG PS 1 | 65 | 128 | 193
Alpha-fetoprotein (AFP) (RAVE) [Count of Participants; unit: Participants] — Alpha-Fetoprotein blood test was performed and baseline data were reported.
  Participants
    less than (<) 400 nanogram per milliliter (ng/mL) | 107 | 217 | 324
    greater than or equal to (>=) 400 ng/mL | 87 | 162 | 249
Alpha-fetoprotein (AFP) (IVRS) [Count of Participants; unit: Participants] — AFP blood test was performed and baseline data were reported.
  Participants
    < 400 ng/mL | 105 | 212 | 317
    >= 400 ng/mL | 89 | 167 | 256
Macrovascular invasion (RAVE) [Count of Participants; unit: Participants] — Macrovascular invasion was defined as presence or absence of invasion of portal or hepatic vasculature by tumor.
  Participants
    Absence | 140 | 269 | 409
    Presence | 54 | 110 | 164
Macrovascular invasion (IVRS) [Count of Participants; unit: Participants] — Macrovascular invasion was defined as presence or absence of invasion of portal or hepatic vasculature by tumor.
  Participants
    Absence | 135 | 262 | 397
    Presence | 59 | 117 | 176
The Barcelona-Clinic Liver Cancer (BCLC) stage at study entry [Count of Participants; unit: Participants] — BCLC classification divides HCC subjects in 5 stages (0=very early stage, A=early stage, B=intermediate stage, C=advanced stage and D=terminal stage) according to pre-established prognostic variables, and allocates therapies according to treatment-related status. Thus, it provides information on both prognostic prediction and treatment allocation.
  Participants
    Early stage | 0 | 1 | 1
    Intermediate stage | 22 | 53 | 75
    Advanced stage | 172 | 325 | 497
Extrahepatic disease (RAVE) [Count of Participants; unit: Participants] — Extrahepatic disease defined as presence or absence of tumor outside the liver.
  Participants
    Absence | 47 | 114 | 161
    Presence | 147 | 265 | 412
Extrahepatic disease (IVRS) [Count of Participants; unit: Participants] — Extrahepatic disease defined as presence or absence of tumor outside the liver.
  Participants
    Absence | 62 | 129 | 191
    Presence | 132 | 250 | 382

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from date of randomization (Day 1) to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From randomization (Day 1) of the first subject until 419 days later
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
days | 237 (192) [192 to 269] | 323 (276) [276 to 369]
Statistical Analysis 1: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio for OS and 95% confidence interval was calculated for stratified IVRS by using Cox model, stratified by the geographic region: Asia or Rest of the World (ROW), ECOG-PS: 0 versus 1, AFP level, presence versus absence of extrahepatic disease and presence versus absence of macrovascular invasion. Kaplan-Meier (KM) estimated for OS and KM survival curves were presented for each treatment arm; Test type: Superiority; p = 0.000017, Log Rank; Hazard Ratio (HR) = 0.624, 95% CI 2-sided [0.498 to 0.782]
Statistical Analysis 2: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio for OS and 95% confidence interval was calculated for stratified RAVE (Sensitivity) by using Cox model, stratified by the geographic region: Asia or Rest of the World (ROW), ECOG-PS: 0 versus 1, AFP level, presence versus absence of extrahepatic disease and presence versus absence of macrovascular invasion. Kaplan-Meier (KM) estimated for OS and KM survival curves were presented for each treatment arm; Test type: Superiority; p = 0.000149, Log Rank; Hazard Ratio (HR) = 0.660, 95% CI 2-sided [0.527 to 0.828]
Statistical Analysis 3: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio for OS and 95% confidence interval was calculated for unstratified (sensitivity) by using Cox model, stratified by the geographic region: Asia or Rest of the World (ROW), ECOG-PS: 0 versus 1, AFP level, presence versus absence of extrahepatic disease and presence versus absence of macrovascular invasion. Kaplan-Meier (KM) estimated for OS and KM survival curves were presented for each treatment arm; Test type: Superiority; p = 0.000107, Log Rank; Hazard Ratio (HR) = 0.674, 95% CI 2-sided [0.546 to 0.831]

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP was the time (days) from randomization to radiological or clinical disease progression assessed by independent radiological review. Median and 95% confidence interval were reported for the modified response evaluation criteria in solid tumors (mRECIST) and response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) analysis sets. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From date of randomization until 30 days after last study treatment (assessed every 6 weeks until PD; and after 8 cycle assessed every 12 weeks) (approximately 33 months)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
days
  mRECIST | 45 (44) [44 to 49] | 97 (87) [87 to 128]
  RECIST 1.1 | 45 (44) [44 to 49] | 119 (87) [87 to 128]
Statistical Analysis 1: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio and its 95% CI was based on stratified (IVRS) Cox Regression Model. One-sided p-value was calculated from log rank test and 95% CIs was computed by using Kaplan-Meier estimates; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.439, 95% CI 2-sided [0.355 to 0.542]
Statistical Analysis 2: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio and its 95% CI was based on unstratified (IVRS) Cox Regression Model. One-sided p-value was calculated from log rank test and 95% CIs was computed by using Kaplan-Meier estimates; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.471, 95% CI 2-sided [0.388 to 0.572]
Statistical Analysis 3: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.412, 95% CI 2-sided [0.334 to 0.509]
Statistical Analysis 4: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.444, 95% CI 2-sided [0.365 to 0.539]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time (days) from date of randomization to date of disease progression (radiological or clinical) or death due to any cause, if death occurs before progression was documented. Death in the absence of progression was a PFS event only if it occurred within the 12+1 weeks for subjects who discontinued treatment prior to cycle 8 and 24+2 weeks for subjects who discontinued treatment after to cycle 8 of the last evaluable tumor assessment; PFS were censored at the date of the last evaluable tumor assessment, if it occurred later. Median and 95% confidence interval 95% were reported for the mRECIST and RECIST 1.1 analysis sets. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From date of randomization until 30 days after last study treatment (assessed every 6 weeks until PD; and after 8 cycle assessed every 12 weeks)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
days
  mRECIST | 45 (44) [44 to 47] | 95 (86) [86 to 127]
  RECIST 1.1 | 45 (44) [44 to 49] | 102 (87) [87 to 127]
Statistical Analysis 1: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio and its 95% CI was based on stratified (IVRS) Cox Regression Model. One-sided p-value was calculated from log rank test and 95% CIs was computed by using Cox Regression Model; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.453, 95% CI 2-sided [0.369 to 0.555]
Statistical Analysis 2: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Hazard ratio and its 95% CI was based on unstratified Cox Regression Model. One-sided p-value was calculated from log rank test and 95% CIs was computed by using Cox Regression Model; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.480, 95% CI 2-sided [0.397 to 0.580]
Statistical Analysis 3: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.347 to 0.522]
Statistical Analysis 4: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.454, 95% CI 2-sided [0.376 to 0.548]

4. Secondary Outcome: Objective Tumor Response Rate (ORR)
Description: Objective tumor response rate (ORR) was defined as the percentage of subjects whose best tumor response CR or Partial Response (PR) observed during trial period assessed according to the mRECIST criteria and RECIST 1.1. CR= Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions. Subjects prematurely discontinuing without an assessment were to be considered non-responders for the analysis.
Time Frame: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
percentage of subjects
  mRECIST | 4.1 | 10.8
  RECIST 1.1 | 2.6 | 6.6
Statistical Analysis 1: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Comparison of treatments were calculated; Test type: Superiority; p = 0.003650, Cochran-Mantel-Haenszel; Difference = -6.88, 95% CI 2-sided [-11.13 to -2.63]
Statistical Analysis 2: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Comparison of treatments were calculated; Test type: Superiority; p = 0.019991, Cochran-Mantel-Haenszel; Difference = -4.15, 95% CI 2-sided [-7.55 to -0.75]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) was defined as the percentage of subjects whose best response was CR (CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target).), PR (PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.), or stable disease (SD) (SD: steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.) according to RECIST and RECIST 1.1 criteria. SD had to be maintained for at least 6 weeks from the first demonstration of that rating.
Time Frame: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
percentage of subjects
  mRECIST | 36.1 | 65.2
  RECIST 1.1 | 34.5 | 65.7
Statistical Analysis 1: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Comparison of treatments were calculated; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Difference = -29.31, 95% CI 2-sided [-37.52 to -21.11]
Statistical Analysis 2: Comparison: Placebo vs Regorafenib 160 mg (BAY73-4506); Comparison of treatments were calculated; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Difference = -31.39, 95% CI 2-sided [-39.57 to -23.22]

6. Other Pre Specified Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from date of randomization (Day 1) to death due to any cause
Time Frame: From randomization (Day 1) of the first subject to end of follow upto 1710 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Regorafenib 160 mg (BAY73-4506)
Number analyzed (Participants) | 194 | 379
days | 241 (196) [196 to 274] | 326 (278) [278 to 372]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after start of study drug administration until 30 days after end of study treatment over a period of approximately three years
Groups:
- Placebo: Description: Subjects received placebo matched to regorafenib tablets orally every day for 3 weeks followed by 1 week off treatment plus best supportive care(BSC).
- Regorafenib (Stivarga, BAY73-4506): Description: Subjects received regorafenib 160 mg (4 *40 mg tablets) orally every day for 3 weeks followed by 1 week off treatment plus BSC.
Arm/Group | Placebo | Regorafenib (Stivarga, BAY73-4506)
All-Cause Mortality (participants affected / at risk) | 176/193 | 324/374
Serious Adverse Events (participants affected / at risk) | 92/193 | 194/374
Other Adverse Events (participants affected / at risk) | 162/193 | 366/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=193) | Regorafenib (Stivarga, BAY73-4506) (N=374)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 4 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (7)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (3)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 6 (7) | 10 (13)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2 (4) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (2) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5) | 6 (6)
Asthenia (General disorders) | 0 (0) | 4 (5)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (3)
General physical health deterioration (General disorders) | 25 (32) | 47 (73)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 6 (6)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (5)
Bile duct stenosis (Hepatobiliary disorders) | 2 (5) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 9 (14) | 9 (14)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatic haemorrhage (Hepatobiliary disorders) | 2 (4) | 2 (3)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (2) | 2 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 2 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (3)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (5)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 4 (5)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Pleural infection bacterial (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 8 (11)
Sepsis (Infections and infestations) | 0 (0) | 3 (5)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (3) | 1 (2)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 2 (3)
Blood pressure decreased (Investigations) | 0 (0) | 1 (2)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (4) | 3 (3)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (6) | 9 (14)
Meningorrhagia (Nervous system disorders) | 0 (0) | 1 (2)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (2)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (2)
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 3 (5)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (3)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (2)
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=193) | Regorafenib (Stivarga, BAY73-4506) (N=374)
Anaemia (Blood and lymphatic system disorders) | 21 (40) | 57 (114)
Hypothyroidism (Endocrine disorders) | 1 (1) | 29 (33)
Abdominal distension (Gastrointestinal disorders) | 10 (13) | 20 (24)
Abdominal pain upper (Gastrointestinal disorders) | 18 (22) | 52 (85)
Abdominal pain (Gastrointestinal disorders) | 29 (43) | 85 (127)
Ascites (Gastrointestinal disorders) | 31 (57) | 61 (91)
Constipation (Gastrointestinal disorders) | 21 (24) | 67 (79)
Diarrhoea (Gastrointestinal disorders) | 31 (44) | 163 (348)
Dry mouth (Gastrointestinal disorders) | 12 (15) | 22 (24)
Nausea (Gastrointestinal disorders) | 26 (38) | 72 (106)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 31 (44)
Vomiting (Gastrointestinal disorders) | 13 (17) | 50 (73)
Asthenia (General disorders) | 19 (34) | 56 (97)
Fatigue (General disorders) | 50 (67) | 110 (205)
Malaise (General disorders) | 5 (5) | 23 (33)
Oedema peripheral (General disorders) | 26 (32) | 63 (81)
Pyrexia (General disorders) | 13 (15) | 79 (113)
Alanine aminotransferase increased (Investigations) | 21 (37) | 56 (102)
Blood alkaline phosphatase increased (Investigations) | 9 (21) | 23 (43)
Aspartate aminotransferase increased (Investigations) | 40 (89) | 99 (234)
Blood bilirubin increased (Investigations) | 30 (59) | 94 (258)
Gamma-glutamyltransferase increased (Investigations) | 14 (32) | 24 (73)
Lipase increased (Investigations) | 7 (15) | 27 (62)
Platelet count decreased (Investigations) | 2 (8) | 39 (129)
Weight decreased (Investigations) | 9 (11) | 55 (132)
Decreased appetite (Metabolism and nutrition disorders) | 29 (37) | 122 (186)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 (19) | 56 (152)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (22) | 28 (62)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (17) | 20 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 15 (17)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (11) | 36 (96)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 50 (73)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (19) | 18 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 38 (48)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 31 (51)
Headache (Nervous system disorders) | 12 (12) | 25 (33)
Insomnia (Psychiatric disorders) | 8 (8) | 30 (35)
Proteinuria (Renal and urinary disorders) | 2 (6) | 34 (96)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 45 (50)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 26 (42)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 68 (85)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 27 (27)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (27) | 194 (554)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (19) | 22 (34)
Rash (Skin and subcutaneous tissue disorders) | 14 (15) | 21 (28)
Hypertension (Vascular disorders) | 14 (30) | 119 (327)
White blood cell count decreased (Investigations) | 2 (7) | 20 (40)

LIMITATIONS AND CAVEATS:
Decimal places were automatically truncated if last decimal equals zero.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less